CLINICAL TRIAL: NCT01741116
Title: A Phase II Study of TKI258 in Patients With Castration-resistant Prostate Cancer
Brief Title: Dovitinib(TKI258) in Patients With Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Kyong-Hwa, Park, Korean Cancer Study Group, Korean Cancer Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-GU11-05; GU11-05 (Other: KCSG)
Record Dates: First submitted 2012-10-17; First posted 2012-12-04 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: castration-resistant prostate cancer; TKI258; FGF23
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TKI258, inhibitor of RTKs (Experimental): Intervention: TKI258
  Investigational drug, TKI258, will be administered to all of the patients after enrollments. Treatment will initially be administered as 28-day cycles as follows:
  - Daily 500mg of TKI258 will be self-administered orally by the patient for 5 days, followed by 2 days of treatment off.
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258 — Investigational treatment refers to TKI258 in this study Until Progression, unacceptable toxicity, withdrawal
  Other Names: Dovitinib

SUMMARY:
The aim of this study is to evaluate efficacy and safety of Dovitinib(TKI258) in patients with castration resistant prostate cancer after failure of docetaxel-based chemotherapy. Further correlative study for metabolic response using PET image and change in serum fibroblast growth factor 23(FGF23) will be conducted.

DETAILED DESCRIPTION:
Growth factor signals are important in carcinogenesis and progression of prostate cancer, and fibroblast growth factors (FGF) have important roles in this regard. FGF ligands (FGF1, -2, -6, -8, and -17) and FGF receptors (FGFR1 and FGFR4) have all shown to be significantly overexpressed in prostate cancer1-5. And, the recent studies have demonstrated that the critical roles of the FGF family members are mediated by the signaling between epithelial and stromal compartments, thus, promoting epithelial-mesenchymal transition (EMT)6,7. Moreover, a recent study has shown that FGF-2 is a mediator of second wave angiogenesis and tumor progression in men during the formation of castration-resistant tumors. Therefore, inhibition of signaling via FGF axis might be a viable strategy for the treatment of castration-resistant prostate cancer.

TKI258, an oral multitargeted receptor tyrosine kinase (RTK) inhibitor is known to potently inhibit the class III, IV, and V RTKs, showing biochemical 50 percent inhibitory concentration(IC50) values <20 nmol/L for VEGFRs (VEGFR-1, VEGFR-2, and VEGFR-3); the platelet-derived growth factor receptor-β (PDGFR-β); fibroblast growth factor receptors 1, 2, and 3 (FGFR-1,2,3); fetal liver tyrosine kinase receptor 3 (FLT-3); and KIT Ret, tyrosine kinase A (TrkA), and csf-1 RTKs. Due to the unique inhibitory activity on FGF pathways, TKI258 has shown significant activity in a variety of tumor xenograft models in athymic mice, including acute myeloid leukemia, multiple myeloma, and colon- and prostate-derived models9.

Castration-resistant prostate cancers (CRPC) are one of the challenges in oncology practice. Although there have been advances in chemotherapy10, new hormonal agents11, and immunotherapeutics12, patients in this subgroup still have limited life expectancy. Therefore, there is an urgent need to identify therapeutic targets and clinical development of target agents for the treatment of CRPC. For this end, sorafenib has been tested in multiple phase II studies earlier13-17; however, the clinical efficacy was very limited. The low efficacy of sorafenib might be partly explained by the lower potency in inhibition of RTKs. Considering nanomolar concentration range of IC50 for TKI258 compared with micromolar concentration for other multi-TKIs, the efficacy of TKI258 should be evaluated in CRPC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed progressive metastatic androgen-independent adenocarcinoma of the prostate with radiographic evidence of disease.
* No more than two previous cytotoxic chemotherapy
* Castration level of testosterone (< 50 ng/dl) achieved by orchiectomy or gonadotropin-releasing hormone(GnRH) agonist
* Eastern Cooperative Oncology Group(ECOG) performance status 0 - 2
* Finished any study drug or chemotherapy earlier than 4 weeks before the first administration of the study drug.
* Age ≥ 20 years old
* Patients must have the following laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 75 x 109/L
  * Hemoglobin (Hgb) > 8 g/dL
  * Serum total bilirubin: ≤ 1.5 x ULN
  * alanine transaminase(ALT) and aspartate aminotransferase(AST) ≤ 2.0 x upper limit of normal(ULN) with or without liver metastases
  * Serum creatinine ≤ 1.5 x ULN or serum creatinine >1.5 - 3 x ULN or 1.5 x ULN<serum creatinine < 3 x ULN, if calculated creatinine clearance (CrCl) is ≥ 30 mL/min using the Cockcroft-Gault equation, see formula below:

CrCl = [140-age (years)] x weight (kg) / [72 x serum Cr (mg/dL)] (if patient is female multiply the above by 0.85)

* Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria

* Patients with known brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases
* Patients with another primary malignancy within 3 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, basal or squamous cell carcinoma or non-melanomatous skin cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
16 week progression free survival rate | Week 16
  disease progression defined as either the appearance of new lesions or unidimensional tumor measurements increasing >20% or symptomatic progression

SECONDARY OUTCOMES:
Overall response rate | up to 24 months
  Overall response rate per Response Evaluation Criteria in Solid Tumors(RECIST)1.0 and Prostate-specific antigen(PSA), overall survival time, toxicity, and biological effect of TKI258 in patients via correlative study using serum and PET-CT image

OTHER OUTCOMES:
Overall survival | up to 36 months
  Overall survival is defined as the time from date of randomization to date of death due to any cause. If the patient is not known to have died, survival will be censored at the date of the last contact. Overall survival will be analyzed at the final analysis cut-off date.
  The Kaplan-Meier product-limit method will be used to describe the overall survival for the study drug (median, 95% confidence intervals, and plots).
Serum FGF23 | 2 months after chemotherapy
  The objective of the exploratory biomarker is to identify a biomarker 'profile' of a patient population most likely to benefit from treatment with TKI258.
  Since this clinical trial was not designed to address specific biomarkers-related hypotheses, the analysis of this data should be viewed as exploratory and hypotheses generating.
PET-CT | 2 months after chemotherapy
  The objective of the exploratory biomarker is to identify a biomarker 'profile' of a patient population most likely to benefit from treatment with TKI258.

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Hwa Park, MD, phD, Principal Investigator — Korea University
Locations (2):
- South Korea (2):
  - Korean Cancer Study Group, Seoul, Chongro-ku
  - Korea University Anam Hospital, Seoul, Seongbuk-gu, Inchon-ro

REFERENCES:
- [Background] Dorkin TJ, Robinson MC, Marsh C, Bjartell A, Neal DE, Leung HY. FGF8 over-expression in prostate cancer is associated with decreased patient survival and persists in androgen independent disease. Oncogene. 1999 Apr 29;18(17):2755-61. doi: 10.1038/sj.onc.1202624. PMID 10348350
- [Background] Gnanapragasam VJ, Robinson MC, Marsh C, Robson CN, Hamdy FC, Leung HY. FGF8 isoform b expression in human prostate cancer. Br J Cancer. 2003 May 6;88(9):1432-8. doi: 10.1038/sj.bjc.6600875. PMID 12778074
- [Background] Heer R, Douglas D, Mathers ME, Robson CN, Leung HY. Fibroblast growth factor 17 is over-expressed in human prostate cancer. J Pathol. 2004 Dec;204(5):578-86. doi: 10.1002/path.1668. PMID 15538740